CLINICAL TRIAL: NCT02982837
Title: Randomized, Multicenter, Open -Label Clinical Trial to Study the Effect of Adding on Pegylated Interferon Therapy for Patients Diagnosed With Chronic Hepatitis B Showing Maintained Response While Receiving Ongoing Nucleotide Analogues
Brief Title: To Study the Effect of Adding on Pegylated Interferon (PEG-INF) Therapy for Patients Diagnosed With Chronic Hepatitis B
Acronym: RC14/055
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: King Abdullah International Medical Research Center (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PDU15001
Record Dates: First submitted 2016-08-07; First posted 2016-12-06 (Estimated); Last update posted 2018-03-09 (Actual); Status verified 2018-01

CONDITIONS: Hepatitis B
MeSH Terms: conditions — Hepatitis B | interventions — Immunomodulation; Nucleosides

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PEG-IFN & NUCLEOTIDE ANALOGUES (Experimental): Peginterferon alfa-2a 180 Mcg infusion per week with ongoing NUCLEOTIDE ANALOGUES for 48 weeks.
  Interventions: Drug: PEG-IFN & Nucleos(t)tide analogues; Drug: Nucleos(t)tide analogues
- NUCLEOTIDE ANALOGUES (Active Comparator): Nucleoside same dose as they started the study.
  Interventions: Drug: Nucleos(t)tide analogues

INTERVENTIONS:
Drug: PEG-IFN & Nucleos(t)tide analogues — Subjects who will be randomized to receive 180 Mcg/ week as an add-on Pegylated Interferon therapy α-2 A with their ongoing NUCLEOTIDE analogues for 48 weeks.
  Other Names: Immunomodulatory therapy
  Arms: PEG-IFN & NUCLEOTIDE ANALOGUES
Drug: Nucleos(t)tide analogues — Subjects will continue on the same dose of Nucleoside/nucleotide analogues as they started the study.
  Other Names: Nucleoside/nucleotide analogues

SUMMARY:
To assess whether PEG-INF (Peglyated - interferon) Add-on therapy in patients of CHB who have achieved a maintained viral suppression (HBV DNA PCR( polymerase chain reaction) <200 for last 3-6 month) with NA's can result in increased rate of HBV infection eradication (HbsAg is undetectable by serological blood testing with or without seroconversion to HBs antibody).

DETAILED DESCRIPTION:
Hepatitis B virus (HBV) infection remains a global health care problem with more than one third of world's population having serological evidence of been exposed to the virus and about 5% of global population ( 350-400 million) being chronically infected. About 15-40% of Patients with chronic hepatitis B (CHB) infection develop complications of liver cirrhosis, liver failure and hepatocellular carcinoma(HCC) in their life time , resulting in an estimated of 500,000 to 1.2 million deaths each year. In Saudi Arabia, chronic hepatitis B remains a serious medical problem, despite the implementation of mandatory HBV vaccination of children since 1989. According to a recent study conducted in Saudi hospital, HBV accounts for 49% of the hepatitis cases . Persistent viral replication is associated with disease progression to liver fibrosis, cirrhosis and development of HCC. Currently two classes of drugs are available for treatment of CHB namely immunomodulatory therapy (conventional & pegylated interferon (Pegasys) PEG-IFN) and nucleoside/nucleotide analogues(NA). Interferon(IFN)-α with its dual immunomodulatory and antiviral effects was the first drug (recombinant standard IFN- α) licensed for Chronic hepatitis B treatment in the 1990's followed by introduction of nucleos(t)ide analogues(NA) in 1998 that directly inhibit HBV polymerase and provide an effective on treatment maintained viral suppression . With the introduction of pegylated interferon- α (PEG-IFN) in 2005 that allows a convenient once a week dosing interval and of equal or superior treatment efficacy than conventional (IFN), the interferon based therapy has markedly improved its utility. Due to its predominant immunomodulatory effect peginterferon (PEG-IFN) offers the advantage of higher sustained off treatment response rate compared to NA thus allowing a finite duration of treatment. The NA act by directly inhibiting HBV polymerase resulting in effective on treatment maintained viral suppression (HBV DNA PCR <200 for last 3-6 month)). However, long term NA therapy has the problems of emergence of viral resistance, long -term safety, cost and patient compliance.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 & < 70 years of both genders.
* CHB on NA's in maintained viral suppression (HBV DNA PCR <200 for last 3-6 month)
* Patients with measurable HBsAg quantitative levels
* Patients with any HBV genotypes.
* Patients with either CHB e Ag positive or eAg negative
* Patients who sign an informed consent for inclusion into the study.
* Patients with hepatitis Delta co-infection.
* only patients with a negative pregnancy test who are of child bearing potential and agree to utilize a strict birth control method will be enrolled

Exclusion Criteria:

* Patients with following characteristics will not be considered for the trial:
* Decompensated liver Cirrhosis
* HCV (hepatitis C virus) or HIV co infection.
* Autoimmune disorders like SLE (Systemic lupus erythematosus), RA (Rheumatoid Arthritis ), AIH (Autoimmune Hemolytic Anemia), ITP (Immune thrombocytopenic purpura), psoriasis etc.
* Untreated psychiatric conditions like depression and alcohol or drug abuse.
* Comorbid conditions like chronic renal failure or post renal/liver transplantation on immunosuppressive therapy.
* Complicated diabetes mellitus and advanced heart failure.
* Pregnancy or not willing to practice contraception.
* Known allergy to Interferons.
* Concomitant treatment with Telbivudine
* Evidence of portal hypertension by Biochemical (Low Platelets less than 100), imaging or UGI (upper gastrointestinal)endoscopy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Estimated)
Dates: Start 2015-03 (Actual); Primary Completion 2019-03 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
The loss of HbsAg between groups (NA) group and NA +Peg_INF group assessed by HbsAg test | 48 weeks
  The loss of HbsAg between groups (NA) group and NA +Peg_INF group assessed by HbsAg test

SECONDARY OUTCOMES:
The seroconversion to HBs antibody between groups (NA) group and NA +Peg_INF group assessed by Hbe Ab test | 6 ,12 months & 48 weeks
  The seroconversion to HBs antibody between groups (NA) group and NA +Peg_INF group assessed by Hbe Ab test
The HBeAg (Hepatitis B e-Antigen) loss in CHRONIC HBV eAg positive patient between groups (NA) group and NA +Peg_INF group assessed by HbeAg test | 6,12 months & 48 weeks
  HBeAg loss in CHRONIC HBV eAg positive patient between groups (NA) group and NA +Peg_INF group assessed by HbeAg test
The conversion of HBeAg to HBe-antibody in CHRONIC HBV eAg (eAntigen) positive patient between groups (NA) group and NA +Peg_INF group assessed by HBe-antibody test | 6,12 months & 48 weeks
  The conversion of HBeAg to HBe-antibody in CHRONIC HBV eAg positive patient between groups (NA) group and NA +Peg_INF group assessed by HBe-antibody test
The correlation between HBsAg ( Hepatitis B Surface Antigen) levels while on therapy at the a defined interval ie 8,12.24,36,48 weeks and rate of HBsAg loss at end of therapy assessed by measuring HBV s Ag during the period 8,12.24,36 and 48 weeks | 8,12,24 and 48 weeks
  The correlation between HBsAg levels while on therapy at the a defined interval ie 8,12.24,36,48 weeks and rate of HBsAg loss at end of therapy assessed by measuring HBV s Ag during that period 8,12.24,36 and 48 weeks
The relationship between HBV genotype and HBsAg loss at the end of the study assessed by measuring HBV genotype only at base line and see if any particular genotype have more HBV sAg loss at the end of the study | At base line & 48 weeks
  The relationship between HBV genotype and HBsAg loss at the end of the study assessed by measuring HBV genotype only at base line and see if any particular genotype have more HBV sAg loss at the end of the study
The relationship between IL28B (Interleukin 28B) genotypes ( polymorphism) and HBsAg loss with or without seroconversion to HBs antibody | At base line & 48 weeks
  The relationship between IL28B genotypes ( polymorphism) and HBsAg loss with or without seroconversion to HBs antibody assess by doing IL28B genotypes ( polymorphism) once during the study and see if any specific IL28B genotypes ( polymorphism) associated more with HBV sAg loss at the end of the study with or without seroconversion to HBs antibody).
The relationship between vitamin D deficiency and (HbsAg loss with or without seroconversion to HBs antibody) assess by measuring Vitamin D level at base line And correlate the baseline level of Vitamin with HBV sAg loss at the end of the study | At base line & 48 weeks
  The relationship between vitamin D deficiency and (HbsAg loss with or without seroconversion to HBs antibody) assess by measuring vitamin D level at base line And correlate the base line level of vitamin D with HBV sAg loss at the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Abduljaleel Alalwan, MD, Principal Investigator — National Guards Health Affairs-Riyadh
Locations (3):
- Saudi Arabia (3):
  - King Abdulaziz Medical City, Jeddah
  - King Abdulaziz Hospital, Jeddah
  - King Abdulaziz Medical City, Riyadh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Goldstein ST, Zhou F, Hadler SC, Bell BP, Mast EE, Margolis HS. A mathematical model to estimate global hepatitis B disease burden and vaccination impact. Int J Epidemiol. 2005 Dec;34(6):1329-39. doi: 10.1093/ije/dyi206. Epub 2005 Oct 25. PMID 16249217
- [Background] Beasley RP. Hepatitis B virus. The major etiology of hepatocellular carcinoma. Cancer. 1988 May 15;61(10):1942-56. doi: 10.1002/1097-0142(19880515)61:103.0.co;2-j. No abstract available. PMID 2834034
- [Background] Bosch FX, Ribes J, Cleries R, Diaz M. Epidemiology of hepatocellular carcinoma. Clin Liver Dis. 2005 May;9(2):191-211, v. doi: 10.1016/j.cld.2004.12.009. PMID 15831268
- [Background] Liaw YF, Chu CM. Hepatitis B virus infection. Lancet. 2009 Feb 14;373(9663):582-92. doi: 10.1016/S0140-6736(09)60207-5. PMID 19217993
- [Background] Al-Tawfiq JA, Anani A. Profile of viral hepatitis A, B, and C in a Saudi Arabian hospital. Med Sci Monit. 2008 Jan;14(1):CR52-56. PMID 18160946
- [Background] Memish ZA, Knawy BA, El-Saed A. Incidence trends of viral hepatitis A, B, and C seropositivity over eight years of surveillance in Saudi Arabia. Int J Infect Dis. 2010 Feb;14(2):e115-20. doi: 10.1016/j.ijid.2009.03.027. Epub 2009 Jun 21. PMID 19540786
- [Background] Chen CJ, Yang HI, Su J, Jen CL, You SL, Lu SN, Huang GT, Iloeje UH; REVEAL-HBV Study Group. Risk of hepatocellular carcinoma across a biological gradient of serum hepatitis B virus DNA level. JAMA. 2006 Jan 4;295(1):65-73. doi: 10.1001/jama.295.1.65. PMID 16391218
- [Background] Chan HL, Tse CH, Mo F, Koh J, Wong VW, Wong GL, Lam Chan S, Yeo W, Sung JJ, Mok TS. High viral load and hepatitis B virus subgenotype ce are associated with increased risk of hepatocellular carcinoma. J Clin Oncol. 2008 Jan 10;26(2):177-82. doi: 10.1200/JCO.2007.13.2043. PMID 18182659
- [Background] Zoulim F, Locarnini S. Hepatitis B virus resistance to nucleos(t)ide analogues. Gastroenterology. 2009 Nov;137(5):1593-608.e1-2. doi: 10.1053/j.gastro.2009.08.063. Epub 2009 Sep 6. PMID 19737565
- [Background] Cooksley WG, Piratvisuth T, Lee SD, Mahachai V, Chao YC, Tanwandee T, Chutaputti A, Chang WY, Zahm FE, Pluck N. Peginterferon alpha-2a (40 kDa): an advance in the treatment of hepatitis B e antigen-positive chronic hepatitis B. J Viral Hepat. 2003 Jul;10(4):298-305. doi: 10.1046/j.1365-2893.2003.00450.x. PMID 12823597
- [Background] Lok AS, McMahon BJ. Chronic hepatitis B. Hepatology. 2007 Feb;45(2):507-39. doi: 10.1002/hep.21513. No abstract available. PMID 17256718
- [Background] Liaw YF, Leung N, Kao JH, Piratvisuth T, Gane E, Han KH, Guan R, Lau GK, Locarnini S; Chronic Hepatitis B Guideline Working Party of the Asian-Pacific Association for the Study of the Liver. Asian-Pacific consensus statement on the management of chronic hepatitis B: a 2008 update. Hepatol Int. 2008 Sep;2(3):263-83. doi: 10.1007/s12072-008-9080-3. Epub 2008 May 10. PMID 19669255
- [Background] Lee A. Prevention of Helicobacter pylori infection. Scand J Gastroenterol Suppl. 1996;215:11-5. PMID 8722377